CLINICAL TRIAL: NCT04724512
Title: Randomised Controlled Trial to Compare Tissue Reactions and Scarring With Polypropylene vs Polyglactin 910 Sutures in Periocular Skin: SUSY Study (SUture StudY)
Brief Title: SUSY Study (SUture StudY) Comparing Scarring With Polypropylene vs Polyglactin 910 Sutures
Acronym: SUSY
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: setup activities were suspended due to COVID
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18SM4898
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Entropion; Inflammation in the Eyelid
MeSH Terms: conditions — Entropion | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: Comparison of different types of stitches to turn the eyelid outwards e.g. polypropylene Vs polyglactin 910 to establish if there is a difference in the level of post-operative inflammation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- polypropylene (Active Comparator): patients randomised to receive polypropylene sutures.
  Interventions: Device: suture
- polyglactin (Active Comparator): patients randomised to receive polyglactin sutures.
  Interventions: Device: suture

INTERVENTIONS:
Device: suture — a type of suture used in entropion surgery

SUMMARY:
Entropion is a common condition in which the ageing eyelid becomes lax and rolls inwards, resulting in the eyelashes rubbing against the surface of the eye. This can cause discomfort, excessive watering and in severe cases inflammation of the surface of the eye which may lead to permanent scarring and impairment of vision.

There are several options for surgical management of entropion. One of the quickest and simplest treatments to turn the eyelid outwards is to have three stitches ('everting sutures') placed into the eyelid. However recurrence of the entropion is common following this procedure alone. A more permanent operation ('definitive surgery') is to shorten and tighten the eyelid ('wedge excision') in addition to the everting sutures. One approach is to perform the everting sutures soon after the patient attends, as this procedure can be done in a clinic or minor operations theatre and provides immediate relief of symptoms, followed by the wedge excision at a later date, when a slot is available in the operating theatre (which has a longer waiting list). These procedures are routinely offered to patients at our hospital.

Different surgeons use different types of stitches to turn the eyelid outwards e.g. polypropylene or polyglactin 910. Currently, there is no consensus as to which stitch causes less inflammation in the eyelid. The aim of this research study is to compare the inflammatory reaction between the two types of stitches. If there is a significant difference, this could provide useful information for surgeons in deciding which stitch is more appropriate for patients, especially those prone to scarring. We will assess the outcome of each type of stitch in terms of objective and clinical assessment of any scars (through questionnaires) and amount of inflammation caused (through examination of the tissue in the lab).

DETAILED DESCRIPTION:
Purpose and design This study will be the first of its kind to address the difference in inflammatory reaction between these two sutures in entropion repair surgery. Both sutures are widely used in the NHS in eyelid surgery already. The study design has involved peer review from eminent doctors and two statisticians. The questionnaire development involved patients.

Recruitment Patients will be recruited from the oculoplastic clinics at the Western Eye Hospital and Royal Bournemouth Hospital where they will be approached by the principal investigator and colleagues who are also members of the regular care team and GCP trained. Patients will be informed about the study and given sufficient time to decide whether or not they wish to participate. Fully informed consent will be obtained before any study procedures will take place.

INCLUSION CRITERIA

* Adult patients (aged 18 years or over)
* Diagnosis of involutional entropion with sufficient lid laxity for a wedge excision
* Ability to provide informed consent EXCLUSION CRITERIA
* Aged under 18 years
* Prior lower eyelid surgery
* Predisposing conditions and treatments known to interfere with scarring and healing

  * Concurrent steroid treatment
  * Addison's disease
  * Poorly controlled diabetes
  * History of keloid scarring
  * History or current cicatrizing disease
  * Warfarin
* Unable to provide informed consent No one will be unfairly excluded/included in the research

Consent Consent will be taken by a researcher who is able to assess capacity and does so in everyday practice. Only participants who are able to give fully informed consent will be approached for participation.

Risks:

The suture material being studied are widely used in oculoplastic surgery internationally and within the NHS. All sutures can cause scarring, although the risk of significant scarring in eyelid surgery is low as eyelids tend to heal well due to a good blood supply. The main risk of surgery is that the procedure does not work, but these are standard NHS treatments and are accepted as being low risk. Patients will be informed that a benefit of being in the trial is that their procedure will be performed by a senior oculoplastic surgeon and much sooner than is usually possible on a standard NHS waiting list. They will have more close attention paid to their symptoms and a more detailed assessment and aftercare.

Confidentiality The investigators will abide by the Caldicott principles. Confidentiality will be maintained at all times in compliance with the ICH GCP and applicable Trust protocols.

Conflict of Interest There is no financial or other conflicts of interest. This is an investigator-led study. Ethicon are providing funding for the study but they have not been involved in the study design and will have no rights over the data handling or publication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or over)
* Diagnosis of involutional entropion with sufficient lid laxity for a wedge excision
* Ability to provide informed consent

Exclusion Criteria:

* Aged under 18 years
* Prior lower eyelid surgery
* Predisposing conditions and treatments known to interfere with scarring and healing

  * Concurrent steroid treatment
  * Addison's disease
  * Poorly controlled diabetes
  * History of keloid scarring
  * History or current cicatrizing disease
  * Warfarin
* Unable to provide informed consent No one will be unfairly excluded/included in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
diameter of the inflammatory reaction around the suture material | 6 months post operation
  The primary outcome measure will be histological, looking at the diameter of the inflammatory reaction around the suture material. In order to minimise the risk of bias from oblique sectioning of the histology, the smallest diameter recorded on each section will be used. Measurements will be taken at 6 levels within the tissue and the mean diameter will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fayers T, Vekinis JS, Ah-Kye L, Parham D, Anketell P, Weir J, A'Hern R, Parkin B. Prospective randomised controlled trial to compare tissue reactions and scarring with polypropylene versus polyglactin 910 sutures in periocular skin. Br J Ophthalmol. 2025 Dec 12:bjo-2025-327724. doi: 10.1136/bjo-2025-327724. Online ahead of print. PMID 41386795